CLINICAL TRIAL: NCT03870906
Title: Assessing the Corporate Environment in Promoting Tobacco Control and Evaluation of a Smoking Cessation Programme in Workplaces in Hong Kong
Brief Title: Smoking Cessation Programme in Workplaces in Hong Kong (Phase IV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Lok Sin Tong Benevolent Society, Kowloon (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LST SCPW P4
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp interaction (Experimental): Individual and group chat interactions.
  Interventions: Behavioral: Occupational-specific health talk; Behavioral: WhatsApp interaction; Behavioral: Phone follow-up/counselling service
- Text message (Placebo Comparator): Regular text messages with similar frequency to those in the Intervention group.
  Interventions: Behavioral: Occupational-specific health talk; Behavioral: Phone follow-up/counselling service; Biological: Text message

INTERVENTIONS:
Behavioral: Occupational-specific health talk — Health talk will provide information about hazards of tobacco (active smoking, second- and third-hand smoke), benefits of quitting smoking and methods to quit smoking.
Behavioral: WhatsApp interaction — Individual WhatsApp interactions last 3-month and consist of 2 parts. First part is regular WhatsApp message. The schedule will be adjusted according to the participants' quitting status. Second part is real-time discussion intervention based on participants' socio-demographic characteristics, smoking habit at baseline and updated smoking status obtained during online conversation. At 3-month follow-up, participants who are still smoking are encouraged to join an additional 1-month online group chat moderated by a smoking cessation counselor.
  Arms: WhatsApp interaction
Behavioral: Phone follow-up/counselling service — The intervention outcomes and participants' smoking status will be followed up regularly via telephone interviews (15 - 30 minutes).
Biological: Text message — Participants will receive regular text messages with similar frequency to those in the intervention group.
  Arms: Text message

SUMMARY:
Smoking causes cardiovascular and respiratory diseases, cancers and diabetes, and it has been a leading risk factor for death globally. Despite the availability of smoking cessation services locally, most smokers do not use such services. Workplace is one of the most convenient platforms to provide smoking cessation services and over 55% of smokers are employed according to the local population-based survey. However, the effectiveness of a smoking cessation programme conducted in workplace is yet to be examined in Hong Kong, and the attitudes and practices of corporations in promoting smoking cessation are not clear. Thus, this study aims to examine the employers'/ managerial staff's knowledge, attitudes and practices in promoting smoking cessation in workplace and evaluate the smoking behaviors of participants before and after attending a smoking cessation intervention.

DETAILED DESCRIPTION:
This study will separate into two phases. Phase I is a large scale cross-sectional survey to corporations in Hong Kong to examine the employers' knowledge, attitudes and practices in promoting smoking cessation in the workplace. Phase II is a 2-arm randomized controlled trial will be conducted to examine the effectiveness of WhatsApp intervention.

Outcome:

The primary outcome of the study is to measure participated smokers' self reported 7-day point prevalence quit rate at 6-month follow-up. Secondary outcomes include participated smokers' (i) self reported 7-day point prevalence quit rate at 9- and 12-month follow-ups; (ii) self-reported reduction rate at 6-, 9- and 12-month follow-ups; (iii) self-reported quit attempt at 6-, 9- and 12-month follow-ups; (iv) change in self-efficacy towards smoking cessation at 6-, 9- and 12-month follow-ups compared with baseline.

Data analyses

Phase I:

Descriptive statistics will be used to measure the (1) basic information of the corporations, including the total number of employees and smoking employees; (2) knowledge on smoking of employers/managerial staff; (3) attitudes on smoking cessation of employers/managerial staff; (4) practices of the corporations with respect to smoking cessation.

Phase II:

Descriptive statistics such as frequency, percentage, and mean will be used to summarize the outcomes and other variables. Chi-square tests and t-tests will be used to compare outcome variables between subgroups. The intention-to-treat analysis will be used such that those lost to contact and refused cases at the follow-ups will be treated as no reduction in cigarette consumption nor quitting. Subgroup analyses will be conducted among the "adherence" cohort, which is classified as subjects who actively participant in the WhatsApp interaction.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least one cigarette per day
* Able to communicate in Cantonese/Mandarin and read Chinese
* Able to use instant messaging tool (e.g. WhatsApp) for communication
* Stay at Hong Kong during the intervention and follow-up periods (12 months)

Exclusion Criteria:

* Smokers who are psychologically or physically unable to communicate
* Currently following other smoking cessation programme(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 6-month
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 9- and 12-month
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up
Self-reported reduction rate | 6-, 9-, and 12-month
  Smokers' who reduced tobacco use (in term of daily cigarette consumption) in the follow-up when comparing with the baseline
Biochemical validation of smoking status | 6-, 9-, and 12-month
  Biochemically validated quit rate (saliva cotinine level and exhale carbon monoxide test)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No